CLINICAL TRIAL: NCT01875055
Title: A Pilot Trial to Assess the Feasibility and Efficacy of Treating Post-Cardiac Surgery Cerebral Desaturation in the Intensive Care Unit
Brief Title: Reversing Cerebral Oxygen Desaturations Greater That 10% of Baseline Values Using NIRS in the ICU
Acronym: NIRS-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B2012:118
Record Dates: First submitted 2013-05-23; First posted 2013-06-11 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2013-02

CONDITIONS: Cerebral Ischemia
Keywords: Cerebral; desaturation
MeSH Terms: conditions — Brain Ischemia | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIRS derived cerebral oximetry (Experimental): NIRS derived cerebral oximetry device used but data not visable to ICU caregivers
  Interventions: Device: NIRS derived cerebral oximetry
- NIRS and Algorithm (Active Comparator): NIRS derived cerebral oximetry device used and the caregiver in the ICU will see the data in order to guide the use of the interventional algorithm to treat the cerebral desaturation
  Interventions: Device: NIRS and Algorithm; Device: NIRS derived cerebral oximetry

INTERVENTIONS:
Device: NIRS and Algorithm — NIRS cerebral oximetry will be used to guide the use of an algorithm based on the modification of previously defined important physiologic variables will be initiated to reverse the desaturation (beginning when the saturation drops at least 10% from the baseline) that occur in the ICU
  Other Names: EQUANOX NIRS derived cerebral oximetry
  Arms: NIRS and Algorithm
Device: NIRS derived cerebral oximetry — NIRS sensors will be placed the forehead of the patient but NIRS derived data will be blinded to the ICU caregivers
  Other Names: EQUANOX NIRS derived cerebral oximetry

SUMMARY:
Study objectives: The main objective of this study is to determine the feasibility of implementing measures in the intensive care unit (ICU), based on a physiological algorithm, to reverse decreases in cerebral oxygen saturation using, near-infrared spectroscopy (NIRS).

Methods: Randomization of 50 patients is balanced by experimental group; control and intervention, with an allocation sequence based on a block size of ten, generated with a computer random number generator. In the intervention group ICU Staff will use NIRS to follow a physiologically guided strategy to maintain regional oxygen saturation (rSO2) within 90% of baseline values. In the control group ICU Staff will provide standard of care without the use of NIRS.

DETAILED DESCRIPTION:
Background and Rationale: Cerebral desaturation has previously been shown to be associated with significant morbidity in cardiac surgery postoperatively. As such, previously reported efforts have been aimed at treating intraoperative desaturation events, with early evidence suggesting that this may reduce the incidence of these adverse events. Our previous study, NIRS ICU (B2011:110) has demonstrated that significant cerebral oxygen desaturation [measured using near infrared spectroscopy (NIRS) derived cerebral oximetry] frequently occurs in the intensive care unit (ICU) within the first 24 hours following cardiac surgery. To date, no studies have addressed the early postoperative period (i.e. in the ICU) with respect to treating (and/or preventing) these desaturation events.

Specific Aims and Experimental Design: The specific aim of this pilot prospective interventional trial is to determine the feasibility/efficacy of treating cerebral oxygen desaturation in the ICU following cardiac surgery. Two groups of patients will be studied. Both groups will have cerebral saturation measured continuously both intraoperatively and postoperatively. The control group however, will have these measurements blinded to the intraoperative and postoperative caregivers. The interventional group will have the cerebral oximetry measurements available to the intraoperative and postoperative care team allowing them to intervene when a desaturation event occurs. If a cerebral desaturation occurs, defined as a decline in saturation of 10% from the patient's preoperative baseline, then a previously utilized interventional algorithm, normal cerebral oxygen saturation (NORMOSAT) (B2012:005), will be instituted to reverse the decrease in cerebral saturation, ideally preventing it from becoming a clinically meaningful desaturation (previously defined by others as saturation decline of 25% from the baseline). The algorithm used addresses many of the known causes of desaturation, including low arterial oxygen content (both saturation and hemoglobin) and cardiac output influences on cerebral blood flow. As such, if a desaturation occurs, the patient will first have the partial pressure of oxygen (PaO2) increased by increasing the inspired oxygen content. The partial pressure of carbon dioxide (PaCO2) will also be normalized by adjusting the ventilator settings. The cardiac output will be optimized and the blood pressure will be increased with standard ICU protocols to administer phenylephrine. If remaining low, the patients will be transfused to standard of care hemoglobin levels.

In this pilot trial, a convenience sample of 50 consecutive consenting patients undergoing cardiac surgery employing cardiopulmonary bypass (CPB) will be studied. After obtaining consent, bilateral cerebral oximetry sensors will be placed on the forehead of patients prior to the induction of anesthesia. Baseline (breathing room air) regional cerebral saturation will be recorded. Following this, induction of anesthesia will occur and continuous NIRS measurements will be collected during the surgical procedure with continued monitoring occurring for the first 24 hours (or until discharge) within the ICU. In the control group, conventional anesthesia and ICU standards of care will be carried out throughout the study period. In the interventional group, an algorithm based on the modification of previously defined important physiologic variables will be initiated to reverse the desaturation (beginning when the saturation drops at least 10% from the baseline) that occurs in the operating room (OR) and ICU.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery employing CPB

Exclusion Criteria:

* patients having surgeries involving the aorta, or employing deep hypothermic circulatory arrest (DHCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence in the two groups of postoperative cerebral desaturation | 24 hours or unit discharge, which ever occurs first.
  Following the end of the 24 hour time period, the NIRS data will be downloaded and analyzed to determine the incidence in the two groups of postoperative cerebral desaturation, primarily defined by a relative reduction in the rSO2 more than 25% from the baseline pre-anesthesia induction. Furthermore, to determine the overall severity of desaturation, the area under the curve (AUC) for a desaturation less than the previously defined 75% of the baseline will be determined. In addition to assessments of endothelial function and delirium, additional patient data on any adverse events will be collected by reviewing the patient charts as well as by phone interview on post-operation day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary P Grocott, MD, Principal Investigator — Professor Department of Anesthesia and Surgery University of Manitoba
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada